CLINICAL TRIAL: NCT02142010
Title: Weekly Paclitaxel Liposome Injection Plus Cisplatin in Preoperative Treatment of Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Luye Sike Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LY-TM-LPS-2014-01
Record Dates: First submitted 2014-05-09; First posted 2014-05-20 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- paclitaxel liposome injection plus cisplatin (Other)
  Interventions: Drug: paclitaxel liposome injection plus cisplatin

INTERVENTIONS:
Drug: paclitaxel liposome injection plus cisplatin — Paclitaxel liposome injection 80 mg/m2, given on days 1, 8,15 and 22 of a 28-day cycle. Cisplatin 25 mg/m2, given on days 1, 8 and 15 of a 28-day cycle, for 4 cycles(4 months)

SUMMARY:
The purpose of this study is to evaluate the pathological complete response (pCR) rate in breast cancer patients treated with weekly paclitaxel liposome injection plus cisplatin preoperative regimen.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥ 18 years and < 65 years,An estimated life expectancy of at least 12 months
* ECOG 0-1
* At least one measurable disease according to the RECIST. histologically confirmed invasive breast cancer, stage II and III, no prior systemic or loco-regional treatment of breast cancer
* Biopsy specimens are available for ER, PgR and Her2 analysis
* Adequate bone marrow function: Neutrophil ≥ 1.5*109/L; Hb ≥ 100g/L; PLT ≥ 100*109/L
* adequate liver function (bilirubin > 1.0 times upper normal limit [UNL] and ALT and/or AST> 1.5 UNL associated with alkaline phosphatase > 2.5 UNL;
* Women with potential child-bearing must have a negative pregnancy test (urine or serum) within 7 days of drug administration and agree to use an acceptable method of birth control to avoid pregnancy for the duration of the study
* No obvious main organs dysfunction
* patients must be accessible for treatment and follow-up and written informed consent

Exclusion Criteria:

* Patient is pregnant or breast feeding
* Inflammatory breast cancer and Metastatic breast cancer
* Patients with medical conditions that indicate intolerant to neoadjuvant therapy and related treatment, including uncontrolled pulmonary disease, diabetes mellitis, severe infection, active peptic ulcer, coagulation disorder, connective tissue disease or myelo-suppressive disease
* History of congestive heart failure, uncontrolled or symptomatic angina pectoris, arrhythmia or myocardial infarction; poorly controlled hypertension (systolic BP > 180 mmHg or diastolic BP > 100 mmHg)
* Has peripheral neuropathy
* Treatment with any investigational drugs within 30 days before the beginning of study treatment
* No psychiatric illness and other situations that would limit compliance of study
* With a history of other malignant tumor
* Known severe hypersensitivity to any drugs in this study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
pathological complete remission (pCR) rate | after 4 months of preoperative treatment

SECONDARY OUTCOMES:
Adverse Events as a Measure of Safety and Tolerability | 4 months during neoadjuvant therapy
clinical response rate | after 4 months of preoperative therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Jiaotong University School of Medicine, Renji Hospital, Shanghai, China